CLINICAL TRIAL: NCT03754049
Title: A Phase 2, Open-label, Pharmacokinetic (PK) Study of a Single Intra-articular Administration of TLC599 in Subjects With Mild to Moderate Osteoarthritis of the Knee
Brief Title: A Phase 2, Open Label, Pharmacokinetic (PK) Study of TLC599 in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLC599A2004
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TLC599 12 mg (Experimental): 12 mg TLC590 (proprietary lipid formulation that consists of 12 mg DSP [active ingredient] with 100 μmol phospholipid) via IA injection in patients with OA of the knee. This 12 mg TLC599 treatment arm consists of six (6) cohorts (G1 to G6), each with different follow-up periods or visit schedules. However, the results will be pooled into a single treatment arm to allow for meaningful analysis across the various synovial fluid (SF) time points, as each subject only has one opportunity to collect an SF sample.
  Interventions: Drug: TLC599
- TLC599 6 mg (Experimental): 6 mg TLC590 (proprietary lipid formulation that consists of 6 mg DSP [active ingredient] with 50 μmol phospholipid) via IA injection in patients with OA of the knee. This 6 mg TLC599 treatment arm consists of two (2) cohorts (G7 and G8), each with different follow-up periods or visit schedules. However, the results will be pooled into a single treatment arm to allow for meaningful analysis across the various synovial fluid (SF) time points, as each subject only has one opportunity to collect an SF sample.
  Interventions: Drug: TLC599
- DSP 4 mg (Active Comparator): Dexamethasone Sodium Phosphate (DSP) at a concentration of 4 mg/mL, 1 mL for a total of 4 mg DSP via IA injection in patients with OA of the knee (G9).
  Interventions: Drug: DSP
- DSP 10 mg (Active Comparator): Dexamethasone Sodium Phosphate (DSP) at a concentration of 4 mg/mL, 2.5 mL for the total of 10 mg DSP via IV injection in healthy subjects (G10).
  Interventions: Drug: DSP

INTERVENTIONS:
Drug: TLC599 — TLC599 is manufactured with the proprietary lipid formulation in lyophilized form (BioSeizer) for the reconstitution with the aqueous DSP (active ingredient).
  Other Names: TLC599 Injection
  Arms: TLC599 12 mg; TLC599 6 mg
Drug: DSP — Dexamethasone sodium phosphate (DSP) is a glucocorticoid widely used in the treatment of joint pain such as gout, osteoarthritis and rheumatoid arthritis via IA injection.
  Other Names: Dexamethasone Sodium Phosphate
  Arms: DSP 10 mg; DSP 4 mg

SUMMARY:
This study is a multi-center, Phase 2, open-label, 1-period, parallel study with 9 cohorts of subjects with osteoarthritis (OA) of the knee enrolled to receive single-dose of TLC599 or Dexamethasone sodium phosphate (DSP) via IA injection and 1 cohort of healthy subjects to receive single-dose of DSP via intravenous (IV) injection.

DETAILED DESCRIPTION:
This Phase 2, open-label, 1 period, parallel study will enroll

1. approximately 90 subjects to receive a single dose of TLC599 or DSP via intra-articular (IA) injection, followed by a PK evaluation period up to 24 weeks and an additional follow-up period of 1 to 5 weeks. Additional subjects may be recruited as needed to achieve at least 10 subjects completing the 1-week blood collection period for each treatment.
2. approximately 12 healthy subjects to receive a single dose of DSP via IV injection, followed by a PK evaluation period up to 1 week and an additional follow-up period of 1 week. Additional subjects may be recruited as needed to achieve at least 12 subjects completing the 48-hour blood collection period for IV DSP.

ELIGIBILITY:
Study Criteria for Patients with OA of the Knee (Cohort G1-G9)

Inclusion Criteria:

* Age 45 or older, non or moderate smokers, body mass index (BMI) ≤ 40.0 kg/m2.
* Knee OA symptoms with confirmed mild to moderate OA.
* Study knee OA severity grade 1-3 (Kellgren-Lawrence).
* Agree to use contraception

Exclusion Criteria:

* Clinically significant (CS) abnormalities (physical, lab, hepatitis B/C, HIV, electrocardiogram [ECG], vital sign or unstable illness).
* Positive urine drug screen, tuberculosis (TB) test; significant alcohol/drug abuse
* Allergic reactions to TLC599, its components, related drugs or cosyntropin.
* History of autoimmune disease, immunodeficiency diseases, treated malignancy, CS opportunistic infection, tuberculosis, infective arthritis or concurrent knee infection
* Intra-articular bleeding in study knee.
* Skin issues at injection site or hindrance to knee joint penetration.
* Blood coagulation disorders.
* Stroke or myocardial infarction
* Poorly controlled hypertension or vital sign abnormalities.
* Interfering conditions with dosing, visits, or compliance or refusal of synovial fluid collection.
* Medication: Strong/moderate Cytochrome P450 (CYP) 3A/3A4 inhibitors/inducers, prescription meds, over-the-counter (OTC)/natural health products, meds affecting platelet function, depot injection/implant, IA corticosteroid, hyaluronic acid, or other injection in study knee, impact on endogenous steroid levels, systemic corticosteroids, live attenuated vaccine, chemotherapeutic/immunosuppressant use for inflammatory diseases.
* Plasma donation or significant blood loss.
* Pregnancy, breastfeeding, or planning to be pregnant/breastfeed
* Serious local/systemic infection or symptomatic viral/bacterial infection
* Severe OA (grade 4) in non-study knee (Kellgren-Lawrence).
* Recent surgery, scheduled knee replacement or lower limb amputation.
* Known/adrenal insufficiency risk.
* Recent participation in other study research

Study Criteria for Healthy Subjects (Cohort G10)

Inclusion Criteria:

* Age 18-45, non-smokers, BMI 18.5-25 kg/m2, body weight ≥ 50.0 kg (males) or ≥ 45.0 kg (females).
* Healthy with no CS illness/surgery within 4 weeks or CS medical history.
* Agree to use contraception
* No new tattoos/body piercings at the injection site until the study ends.

Exclusion Criteria:

* CS abnormal physical, ECG or vital sign findings.
* Known/adrenal insufficiency risk.
* Abnormal lab results (HBV, HCV, HIV, TB).
* Positive pregnancy test or lactating; positive urine drug screen or cotinine test.
* Significant alcohol/drug abuse or positive alcohol test.
* Significant drug allergies or allergic reactions to DSP, dexamethasone, cosyntropin, natural adrenocorticotropic hormone (ACTH), or other related drugs.
* History/presence of conditions including CS opportunistic infection, serious local/systemic infection, autoimmune, blood, heart, vascular, respiratory, lung, skin, liver, gallbladder, retinopathy, neuromuscular, cancer, kidney, diabetes, severe allergic reactions, or others that would preclude participation.
* Fever
* Active/latent tuberculosis or symptomatic viral/bacterial infection
* Medication: Depot injection/implant, vaccine, drug known to induce or inhibit CYP3A4 metabolism, prescription meds, OTC/natural health products.
* Consumption of specified fruits.
* Recent participation in other study research
* Plasma donation or significant blood loss.
* Reasons preventing study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Area under the Curve [AUC] | Baseline till 24 weeks post investigational product (IP) administration
  Area under the concentration-time curve
Cmax: maximum concentration | Baseline till 24 weeks post IP administration
  Maximum concentration
Tmax: time to peak concentration | Baseline till 24 weeks post IP administration
  Time to peak concentration

SECONDARY OUTCOMES:
Number of adverse events (AEs), including serious adverse event (SAE) and treatment-emergent AE | Screening till 25 weeks post IP administration
  Number of AEs, including SAE and treatment-emergent AE
Cortisol concentration | baseline till 24 weeks post IP administration
  Cortisol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Terry Tai, MD, Study Director — Taiwan Liposome Company
Locations (10):
- United States (7):
  - Arizona Research Center, Phoenix, Arizona
  - Panax Clinical Research, Miami, Florida
  - South Coast Research Center, Miami, Florida
  - Syneos Health, Miami, Florida
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Futuro Clinical Trials, LLC., McAllen, Texas
  - JBR Clinical Research, Salt Lake City, Utah
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No